CLINICAL TRIAL: NCT01484600
Title: Study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of REGN668 Administered Subcutaneously to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R668-HV-1108
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental)
  Interventions: Drug: REGN668: Injection Rate 1
- Group 2 (Experimental)
  Interventions: Drug: REGN668: Injection Rate 2

INTERVENTIONS:
Drug: REGN668: Injection Rate 1 — Subjects will receive REGN668 via SC injection
  Arms: Group 1
Drug: REGN668: Injection Rate 2 — Subjects will receive study drug via alternate delivery (if necessary)
  Arms: Group 2

SUMMARY:
This is a study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of REGN668 Administered Subcutaneously to Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 55 years of age.
2. Body weight between 60 kg and 80 kg, body mass index between 20 and 30 kg/m2 inclusive.
3. NHV as evidenced by comprehensive clinical assessment (detailed medical history and complete physical examination).
4. Normal resting blood pressure and heart rate
5. Willingness to refrain from the consumption of alcohol for 24 hours prior to each study visit.

Exclusion Criteria:

1. History or presence of currently relevant medical conditions, including any cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, musculoskeletal, psychiatric, systemic, ocular, infectious or parasitic disease, or signs of acute illness.
2. Administration of any medications within 1 week before randomization, other than vitamins, nutritional supplements, or low doses of aspirin taken prophylactically.
3. Onset of a new exercise routine or major change to a previous exercise routine within 2 weeks prior to randomization. Subjects must be willing to maintain a relatively constant level of exercise during the study and refrain from unusually strenuous physical activities
4. Known history of human immunodeficiency virus (HIV) antibody; and/or positive hepatitis B surface antigen (HBsAg), and/or positive hepatitis C antibody (HCV) at the screening visit.
5. History of substance (eg. drug or alcohol) abuse or regular (daily) smoking within a year prior to randomization or positive results on urine drug screen.
6. Excessive consumption of beverages with xanthine derivates (caffeine, theophylline, theobromine), such as coffee, tea, cola, or yerba mate (more than 4 cups or glasses per day).
7. Hospitalization for any reason within 60 days of randomization.
8. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days of the investigational drug, whichever is longer, prior to the randomization visit.
9. Live/attenuated vaccinations within 12 weeks of randomization or during the study.
10. Tuberculosis vaccination within the last year.
11. Previous exposure to any other biological agent within 12 months of randomization.
12. History of a hypersensitivity reaction to doxycycline or other tetracyclines.
13. Recent travel (within 12 months of randomization) to areas endemic for parasitic helminthes, such as developing countries, particularly in Africa and the tropical and subtropical regions of Asia.
14. Pregnant or breast-feeding women.
15. Unwilling to use adequate birth control if of reproductive potential and sexually active

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Baseline through day 64 (end of study)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile of REGN668 | Baseline through day 64
Incidence of anti-REGN668 antibodies | Day 29 and Day 64

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- San Antonio, Texas, United States

REFERENCES:
- [Derived] Li Z, Radin A, Li M, Hamilton JD, Kajiwara M, Davis JD, Takahashi Y, Hasegawa S, Ming JE, DiCioccio AT, Li Y, Kovalenko P, Lu Q, Ortemann-Renon C, Ardeleanu M, Swanson BN. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Dupilumab in Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2020 Aug;9(6):742-755. doi: 10.1002/cpdd.798. Epub 2020 Apr 29. PMID 32348036